CLINICAL TRIAL: NCT05313022
Title: A Randomized, Double-blinded, Placebo-controlled Clinical Trial to Evaluate the Immunogenicity and Safety of the Recombinant SARS-CoV-2 Vaccine (CHO Cell) in Healthy Adults Aged 60 Years and Above
Brief Title: Safety and Immunogenicity of Recombinant SARS-CoV-2 Spike Protein Vaccine (CHO Cell) for the Prevention of COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Collaborators: Walvax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202-COV-1003
Record Dates: First submitted 2022-03-05; First posted 2022-04-06 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ZR-202-CoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZR-202-CoV (Experimental): Adult healthy subjects (60 years of age above, inclusive) receive ZR-202-CoV at Day 0 and Day 28
  Interventions: Biological: ZR-202-CoV
- Placebo (Placebo Comparator): Adult healthy subjects (60 years of age and above) receive 2 doses of placebo (saline) at Day 0 and Day 28
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ZR-202-CoV — Adjuvanted Recombinant SARS-CoV-2 S-protein Subunit Vaccine
  Arms: ZR-202-CoV
Other: Placebo — Normal saline solution
  Arms: Placebo

SUMMARY:
The purpose of this double-blind, randomized, controlled study is to assess safety, reactogenicity, and immunogenicity of ZR-202-CoV, administered as 2 injections (i.m) at 28 days apart in adult subjects 60 years of age and above.

ELIGIBILITY:
Inclusion Criteria:

* Having understood the contents of the clinical study and ICF, and having signed the ICF.
* Adults of both genders, 60 years of age and older.
* Adults who can provide legal proof of identity.
* SARS-COV-2 antibody screening negative at screening visit.

Exclusion Criteria:

* Having a clear or suspected allergy to the test vaccine ingredients (including S protein, aluminum hydroxide adjuvant or CpG adjuvant), or have a history of severe allergy to any previous vaccine (such as acute allergic reaction, dyspnea or angioneurotic edema, etc.) (inquiries);
* Having a history of SARS or MERS infection, or a previous infection of COVID-19 (previous nucleic acid or serum antibody test was positive) (inquiries);
* Previous vaccination with SARS-CoV-2 vaccine(including SARS-CoV-2 vaccine for clinical trial) or received other vaccines within 28 days prior to the first dose of vaccine;
* Abnormal skin (such as inflammation, induration, redness and swelling, large area scar, etc.) on both sides of the arm at the vaccination site and affecting the vaccination or safety observation(examination);
* Axillary body temperature ≥37.3℃ before the first dose vaccination(examination);
* Safety laboratory abnormal of any of the below:

  1. Liver function: ALT or ALT > 1.25*ULN
  2. Kidney function: serum creatinine (Cr) > ULN
  3. Glycated hemoglobin (HbA1c) ≥ 8.0%
* Uncontrolled epilepsy or other progressive neurological diseases (inquiries);
* Immunocompromised or have been diagnosed with Human Immunodeficiency Virus (HIV) infection, lymphoma, leukemia, Systemic lupus erythematosus, SLE, rheumatoid arthritis, inflammatory bowel disease or other autoimmune diseases (inquiries);
* Asplenia or functional asplenia (inquiries);
* Having a history of coagulation disorder or abnormal coagulation function (e.g., lack of coagulation factors or thrombocytopenia) and assessed by investigators that are not suitable for the study (inquiry);
* Having malignant tumor that not been cured clinically and been assessed by investigators as not suitable for the study (inquiry);
* Having acute diseases or acute onset or poorly controlled chronic diseases(e.g. hypertension patients with blood pressure > 160/100mmHg, diabetes patients with ketoacidosis, etc.) within 14 days before the first dose vaccination and assessed by investigators as not suitable for the study (inquiry);
* Use of systemic drugs that affect immune function within 6 months prior to the first dose vaccination for a long time (more than 14 consecutive days), such as immunosuppressant, cytotoxic drugs, inhaled corticosteroids (not including allergic rhinitis treated with corticosteroid spray), unless the investigators determines that the drug will not interfere with, limit, or obfuscate the evaluation prescribed by the protocol, or may endanger the safety of the subject (inquiry);
* Treatment with whole blood, plasma or immunoglobulin within 3 months prior to the first dose(inquiry);
* Any other factors that, in the investigator's judgment, are inappropriate for participation in the clinical study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 neutralising antibody | 28 days after each dose
Proportion of participants achieving seroconversion for SARS-CoV-2 neutralising antibody | 28 days after each dose
Geometric mean increase (GMI) of SARS-CoV-2 neutralising antibodies | 28 days after each dose
Geometric mean titer (GMT) of SARS-CoV-2 specific IgG binding antibodies. | 28 days after each dose
Proportion of participants achieving seroconversion for SARS-CoV-2 specific IgG binding antibodies.. | 28 days after each dose
Geometric mean increase (GMI) of SARS-CoV-2 specific IgG binding antibodies. | 28 days after each dose

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) after vaccination | 28 days after the first or second vaccination
  Percentage of participants with AEs for 28 days following each vaccination (Days 0, 28) by intensity, relevance.
Incidence of solicited adverse events (AEs) after vaccination | 30 minutes and 7 days after the first or second vaccination
  Percentage of participants with solicited AEs for 30 minutes and 7 days following each vaccination (Days 0, 28) by intensity, relevance
Incidence of unsolicited adverse events (AEs) after vaccination | 28 days after the first or second vaccination
  Percentage of participants with unsolicited AEs for 28 days following each vaccination (Days 0, 28) by intensity, relevance.
Proportion of subjects with abnormal markers of hematology, biochemistry, urinalysis, thyroid and coagulation parameters | Day 4 after first or second vaccination
  Safety Laboratory Values (Serum Chemistry, Hematology)
Incidence of serious AEs (SAEs) and adverse events of special interest (AESIs) | up to 12month after last dose vaccination
  Percentage of participants with SAEs or AESIs for 12month after last dose vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Institution for Anning First Hospital, Kunming, Yunan, China